CLINICAL TRIAL: NCT05604781
Title: Evaluating A Novel Strategy: The Synergy IOL Mixed and Matched With the Symfony With Intelilight
Brief Title: Symfony/Synergy IOL Combination Outcomes
Status: Completed | Type: Observational
Sponsor: Center For Sight (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Other Study IDs: CFS-22-001
Record Dates: First submitted 2022-10-26; First posted 2022-11-03 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Bilateral Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Symfony & Synergy IOL combination
  Interventions: Device: Symfony & Synergy IOL combination

INTERVENTIONS:
Device: Symfony & Synergy IOL combination — The Symfony IOL will be implanted in the dominant eye while the Synergy IOL will be implanted in the non-dominant eye.

SUMMARY:
Current visual outcomes expectations of cataract patients are similar to those of refractive surgery patients. Their desire is to be spectacle independent for far, intermediate and near vision activities. Some may have already enjoyed freedom from glasses and would like to continue after the cataracts are removed. Different options are available. These options include: mono-vision and presbyopia correcting intraocular lenses (IOL). Presbyopia correcting IOLs include accommodative, multifocals and extended depth of focus (EDOF) IOLs. In a previous study that evaluated the visual outcomes of an EDOF IOL when combined with a multifocal IOL with a +3.25 D add in patients with or without astigmatism undergoing routine cataract surgery showed good outcomes with high patient satisfaction and less dependance on glasses for intermediate and near activities. As technology evolves, new lens models are available in the market. The purpose of this study is to evaluate the latest EDOF and a hybrid multifocal lenses when combined.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing bilateral lens extraction with intraocular lens implantation of the Symfony with InteliLight in the dominant eye and a Synergy in the non-dominant eye.
2. Gender: Males and Females.
3. Age: 50 years and older.
4. Willing and able to provide written informed consent for participation in the study
5. Willing and able to comply with scheduled visits and other study procedures.
6. Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 2 to 30 days between surgeries
7. Subjects who require an IOL power in the range of +5.00 D to +34.0 D only.
8. Subjects who require a toric IOL up to +3.75 D at the IOL plane (2.57 D corneal plane).
9. Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

1. Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
2. Uncontrolled diabetes.
3. Use of any systemic or topical drug known to interfere with visual performance.
4. Contact lens use during the active treatment portion of the trial.
5. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
6. Clinically significant corneal dystrophy
7. History of chronic intraocular inflammation.
8. History of retinal detachment.
9. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
10. Previous intraocular surgery.
11. Previous corneal refractive surgery (i.e. LASIK, photorefractive keratectomy, radial keratotomy).
12. Previous keratoplasty
13. Severe dry eye
14. Pupil abnormalities
15. Anesthesia other than topical or peribulbar anesthesia (i.e. retrobulbar, general, etc).
16. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
17. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from two ophthalmology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center For Sight, Venice, Florida
  - Helga Sandoval, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soscia WL, DeRojas JO, Mathews PM, Brutsky A, Solomon KD, Potvin R, Sandoval HP. Clinical performance after implantation of an EDOF intraocular lens in the dominant eye and a presbyopia-correcting intraocular lens in the nondominant eye. J Cataract Refract Surg. 2024 Jun 1;50(6):578-584. doi: 10.1097/j.jcrs.0000000000001412. PMID 38305420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symfony & Synergy IOL Combination
Started | 41
Completed | 37
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Symfony & Synergy IOL Combination
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Binocular Defocus Curve
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Symfony & Synergy IOL Combination
Number analyzed (Participants) | 37
logMAR
  +1.00 D | 0.07 (0.10)
  +0.50 D | -0.05 (0.08)
  0.00 D | -0.08 (0.12)
  -0.50 D | -0.05 (0.09)
  -1.00 D | -0.04 (0.10)
  -1.50 D | -0.03 (0.13)
  -2.00 D | 0.04 (0.13)
  -2.50 D | 0.07 (0.14)
  -3.00 D | 0.14 (0.14)

2. Secondary Outcome: Patient Satisfaction Questionnaire
Description: Percentage for participants who are completely or mostly satisfied with their overall vision will be assessed
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Symfony & Synergy IOL Combination
Number analyzed (Participants) | 37
Participants | 31

3. Secondary Outcome: Spectacle Independence for Near Activities Questionnaire
Description: Percentage of participants reporting the need to wear glasses all the time for near activities will be assessed.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Symfony & Synergy IOL Combination
Number analyzed (Participants) | 37
Participants | 4

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Symfony & Synergy IOL Combination
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT05604781/Prot_SAP_000.pdf